CLINICAL TRIAL: NCT05494476
Title: Stability of the Marginal Bone Around Subcrestal Implants Inserted at Different Depths. A Multicenter Clinical Study
Brief Title: Stability of the Marginal Bone Around Subcrestal Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MEGADEPTH
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Alveolar Bone Loss; Dental Implant Failure Nos
Keywords: marginal bone loss; peri-implant bone remodeling; submerged dental implant
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: split mouth protocol
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2mm under bone level (Active Comparator): implant platform will be submerged 2mm under bone level
  Interventions: Procedure: implant insertion
- 1mm under bone level (Active Comparator): implant platform will be submerged 1mm under bone level
  Interventions: Procedure: implant insertion

INTERVENTIONS:
Procedure: implant insertion — after flap detachment, implant bed will be prepared with twist-drill, implant will be inserted according to randomization (1 or 2 mm under bone)

SUMMARY:
The extent of marginal bone remodeling around the neck of dental implants has been used for many years as a criterion for defining their long-term success. Apico-coronal position represents a crucial factor in this field. This study aims to establish the optimal insertion depth of a subcrestal implant, with the aim of minimizing the bone resorption.

DETAILED DESCRIPTION:
The extent of marginal bone remodeling around the neck of dental implants has been used for many years as a criterion for defining their long-term success.

In reality, the etiology of this bone remodeling (Marginal Bone Loss-MBL) has not yet been well understood, although many theories have been proposed to explain it.

The influence of mucosal thickness on marginal bone loss has been discussed by Cochran et al., which suggest a protective action for the underlying soft tissue bone that recreates a sort of "biological width" around the implant. In fact, some studies have hypothesized that a marginal bone loss> 2.0 mm provides the vertical space for the correct restoration of biological width. Linkevicius et al. have published various studies that have shown that, in crestally placed implants with switching platform, a vertical thickness of the soft tissues greater than 2 mm is effective in preventing the loss of peri-implant marginal bone. However, other authors have demonstrated significant marginal bone loss around implants with low prosthetic abutments compared to those with higher prosthetic abutments. In particular, the extent of bone loss was more reduced when the height of the abutment was> 2 mm. From a theoretical point of view, a 3 mm high prosthetic abutment, calculated from the apical edge of the crown to the implant platform, should provide adequate space for restoring biological width.

Furthermore, a recent study conducted on subcrestal implants has shown that early marginal bone resorption, in addition to being linked to the thickness of the soft tissues and the height of the abutment, is negatively influenced by the depth of implant insertion. However, the same study underlines that implants inserted more deeply, while losing more marginal bone than more superficial implants, are covered by a greater bone thickness at the end of the remodeling process.

This study aims to establish the optimal insertion depth of a subcrestal implant, with the aim of minimizing the resorption of the marginal bone and keeping the implant platform below the bone level after 12 months of prosthetic loading.

ELIGIBILITY:
Inclusion Criteria:

* indications for the insertion of two implants in a free edentulous ridge in the posterior area of both arches (premolar / molar area), based on a careful diagnosis and treatment plan;
* presence of a residual bone crest with a minimum surgical height of 9 mm, and a thickness of at least 6 mm at the level of the planned implant sites;
* the bone crest must be healed (at least 6 months after tooth loss / extraction of the corresponding dental element);
* native bone;
* plaque index below 25% and bleeding index below 20%;
* facial-lingual width of the adherent gingiva ≥ 4 mm;
* age of the patient> 18 years;
* patients must be able to review and understand the study protocol;
* informed consent.

Exclusion Criteria:

* acute myocardial infarction within the last 6 months;
* uncompensated coagulation disorders;
* uncontrolled diabetes (HbA1c> 7.5%);
* head / neck radiotherapy in the last 24 months;
* immunocompromised patients (HIV infection or chemotherapy within the last 5 years);
* present or past treatment with antiresorptive drugs;
* psychological or psychiatric problems;
* alcohol or drug abuse;
* presence of uncontrolled periodontal disease
* acute and chronic endodontic infections next to implant site.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
marginal bone loss | at implant insertion
  radiographic assessment
marginal bone loss | 5 month after implant insertion
  radiographic assessment
marginal bone loss | 6 months after prosthetic loading
  radiographic assessment
marginal bone loss | 12 months after prosthetic loading
  radiographic assessment
marginal bone loss | 3 years after prosthetic loading
  radiographic assessment
marginal bone loss | 5 years after prosthetic loading
  radiographic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr, Study Director — Piezoelectric Surgery Academy
Locations (1):
- Dr. Claudio Stacchi Office, Gorizia, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spinato S, Stacchi C, Lombardi T, Bernardello F, Messina M, Zaffe D. Biological width establishment around dental implants is influenced by abutment height irrespective of vertical mucosal thickness: A cluster randomized controlled trial. Clin Oral Implants Res. 2019 Jul;30(7):649-659. doi: 10.1111/clr.13450. Epub 2019 May 12. PMID 31033035
- [Background] Galindo-Moreno P, Leon-Cano A, Monje A, Ortega-Oller I, O'Valle F, Catena A. Abutment height influences the effect of platform switching on peri-implant marginal bone loss. Clin Oral Implants Res. 2016 Feb;27(2):167-73. doi: 10.1111/clr.12554. Epub 2015 Feb 11. PMID 25678247